CLINICAL TRIAL: NCT06171139
Title: Developing and Testing a Patient-centered Tumor Genomic Pre-test Counseling Tool for Black or African-American Men With Metastatic Prostate Cancer
Brief Title: Tumor Genomic Pre-test Counseling Tool for Black or African-American Men With Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23553; NCI-2023-10339 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1: Tool Development (Experimental): Participants will participate in a semi-structured qualitative interview either by phone, video conference or in-person. A trained interviewer will interview eligible, consenting participants using a semi-structured interview guide to meet objectives. The interview guide is based on The Patient Education Materials Assessment Tool (PEMAT) and the COM-B (capability (C), opportunity (O), and motivation (M))/Behaviour Change Wheel (BCW) framework and will be used to determine an implementation strategy. The interview will be audio-recorded, transcribed verbatim, and analyzed.
  Interventions: Other: Counseling Tool; Other: Questionnaires
- Stage 1: Tool Implementation (Pilot Study) (Experimental): Participants will receive the tumor genetic pre-test counseling tool informed by results and themes identified in Stage 1. Participants will receive the non-therapeutic intervention, a pre-TGT counseling tool, and complete pre- and post-intervention surveys and a attend a brief post-intervention interview.
  Interventions: Other: Counseling Tool; Other: Questionnaires

INTERVENTIONS:
Other: Counseling Tool — Non-therapeutic educational intervention
Other: Questionnaires — Participants will complete questionnaires online, via mail, by telephone, or in person per participant preference.
  Other Names: Surveys

SUMMARY:
The overall goal of the study is to improve equitable delivery of pre-Tumor genetic testing (TGT) counseling tool for Black or African American men with metastatic prostate cancer and evaluating the tool for implementation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Stage 1: To evaluate education quality of the intervention in Black or African American men with prostate cancer.

Stage 2: To evaluate feasibility of the TGT intervention among Black or African American men with prostate cancer

SECONDARY OBJECTIVES:

Stage 1:

1. To evaluate completeness of the intervention content.
2. To identify barriers and facilitators for using the intervention.

Stage 2:

1. To evaluate the acceptability of the intervention among Black or African American men with prostate cancer.
2. To evaluate change in participant knowledge about tumor genetic testing among Black or African American men with prostate cancer.
3. To evaluate change in patient attitudes toward tumor genetic testing among Black or African American men with prostate cancer.
4. To evaluate change in participant expectations of tumor genetic testing among Black or African American men with prostate cancer.
5. To evaluate patient perspectives on the intervention.
6. To evaluate the rate of TGT among Black or African American men with prostate cancer who have received the tumor genetic pre-test counseling tool.

OUTLINE:

This is a two-stage study. In Stage 1, Adult Black or African American men with metastatic prostate cancer who have not made a decision about TGT, or who have decided to undergo TGT, or patients who have decline TGT about tumor genetic testing will participate in development by answering questionnaires and utilizing the pilot application for up to 60 days. The investigators will then refine the tool to be piloted in Stage 2.

Stage 2: A pilot study of participants who are planning to have a discussion about undergoing tumor genetic testing with their oncology provider will be invited to join and utilize the tool, and answer questionnaires about the tool.

ELIGIBILITY:
Inclusion Criteria:

Stage 1:

1. Age 18-years-old or older
2. Identifies as Black or African American, by either chart documentation or participant self-report. Mixed-race including Black or African American is included.
3. Metastatic prostate cancer, by either chart documentation or participant self-report. Pathology report not needed.
4. Able to understand study procedures and to comply with them for the entire length of the study.
5. Able to understand a written information sheet and willing to verbally consent.
6. Fluent in English (reading, writing, and speaking)

Stage 2:

1. Age 18-years-old or older
2. Identifies as Black or African-American, by either chart documentation or participant self-report. Mixed-race including Black or African-American is included.
3. Metastatic prostate cancer, by either chart documentation or participant self-report. Pathology report not needed.
4. Able to understand study procedures and to comply with them for the entire length of the study.
5. Fluent in English (reading, writing, and speaking).
6. Anticipated discussion of TGT within 0-90 days of enrollment, per treating oncology provider's discretion. TGT involves use of any cancer genetic sequencing (whether standard-of-care or part of a research protocol) via any one of the following:

   1. Somatic DNA testing of already-collected tissue.
   2. Somatic DNA testing of tissue to be collected in the future via biopsy, surgery, or other procedure.
   3. Blood-based DNA testing to evaluate for circulating tumor DNA.
7. Able to understand a written informed consent document and willing to sign it.

Exclusion Criteria:

Contraindication to any study-related procedure or assessment in either stage.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of participant responses (Stage 1) | 1 day
  Participant-reported perspectives of intervention in a semi-structured interview will be collected during Stage 1 and reviewed and will be explored using thematic analysis. A codebook will be created using the PEMAT (for the primary objective) described in the interview guide. This framework provides a systematic approach for identifying behavior change models evaluated according to three criteria: comprehensiveness, coherence, and a clear link to an overarching model of behavior. This will produce evidence-based behavior change techniques most likely to be effective. Emergent codes and themes will be added throughout thematic analysis. Two coders will code each interview (one primary and one secondary coder). Discrepancies will be negotiated to consensus.
Proportion of enrolled participants (Stage 2) | 1 day
  The proportion of participants who enrolled in the study after being approached by their healthcare team will be reported.
Proportion of enrolled participants who review all educational materials (Stage 2) | Up to 60 days
  The proportion of all enrolled participants who utilized and reviewed all of the educational materials in the tool will be reported.
Mean score of Feasibility of Intervention Measure (FIM) (Stage 2) | Up to 60 days
  Scores on the FIM will be averaged across all participants. Items will be scored on a 5-point scale: 1= Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5= Completely agree. A higher mean score indicates greater feasibility. The mean score and standard deviation will be reported.

SECONDARY OUTCOMES:
Mean score of Acceptability of Intervention Measure (AIM) (Stage 2) | Up to 60 days
  Scores on the AIM items will be averaged across all participants. Items will be scored on a 5-point scale: 1= Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5= Completely agree. A higher mean score indicates greater feasibility. The mean score and standard deviation will be reported.
Mean score of investigator-developed, measure of acceptability items (Stage 2) | Up to 60 days
  Scores on the 5-item investigator-developed, measure of acceptability will be scored on a 5-point scale: 1= Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5= Completely agree. A higher mean score indicates greater feasibility. The mean score and standard deviation will be reported. However, responses will not be averaged to across items; each item will be analyzed independently.
Mean score of cancer genomic testing knowledge (Stage 2) | Up to 60 days
  Knowledge of tumor genetic testing adapted from a validated survey from Blanchette, et al.+ select questions from a survey from Rogith, et al.will be utilized to measure the level of cancer genomic testing knowledge. "Don't know" will be scored as incorrect. The proportion of correct responses will be calculated to generate a total score between 0-100, with a higher score indicating greater knowledge. No items will be weighted. Since all items are required, we anticipate missing responses will be rare. Any missing data will be managed case-by-case post-hoc.
Proportion of participants who select correct response in each genomic testing knowledge instrument item (Stage 2) | Up to 60 days
  Knowledge of tumor genetic testing adapted from a validated survey from Blanchette, et al. including select questions from a survey from Rogith, et al. and is designed to measure the level of cancer genomic testing knowledge. Responses of "Don't know" will be scored as incorrect. Each of the item scores will be reported as a proportion of the participants who answered each item correctly. Since all items are required, we anticipate missing responses will be rare. Any missing data will be managed case-by-case post-hoc.
Proportion of participants who answer "Yes" to each attitude item in the Attitude and expectations for tumor genetic testing survey (Stage 2) | Up to 60 days
  Attitude and expectations measure for tumor genetic testing is a 17-item measure adapted from a validated survey from Blanchette, et al. including one open-ended investigator-created item. Items on the attitude scoring scale range from "Yes" = 1 and "No" or "Unsure" = 0.
Proportion of participants who answer "Strongly Agree" or "Agree" to the expectation item in the Attitude and expectations for tumor genetic testing survey (Stage 2) | Up to 60 days
  The attitude and expectations for tumor genetic testing is a measure adapted from a validated survey from Blanchette, et al. and includes one open-ended investigator-created item. The expectations scoring (item 3): "Strongly Agree" or "Agree" = 1 and all other responses = 0
Participant-reported perspectives of intervention in a semi-structured interview. (Stage 2) | Up to 60 days
  Participant-reported perspectives of intervention in a semi-structured interview will be collected during Stage 1 and reviewed and will be explored using thematic analysis. A codebook will be created using the COM-B ((capability (C), opportunity (O), and motivation (M) / BCW domains (for the secondary objectives) described in the interview guide. This framework provides a systematic approach for identifying behavior change models evaluated according to three criteria: comprehensiveness, coherence, and a clear link to an overarching model of behavior. This will produce evidence-based behavior change techniques most likely to be effective. Emergent codes and themes will be added throughout thematic analysis. Two coders will code each interview (one primary and one secondary coder). Discrepancies will be negotiated to consensus.
Proportion of participants who have received the tumor genetic pre-test counseling tool who undergo TGT by chart review (Stage 2) | Up to 90 days
  A medical record review of TGT completion date will be conducted. If TGT was not completed, the study staff will review and record reasons for non-completion, and date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kwon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No